CLINICAL TRIAL: NCT05422625
Title: Percutaneous Tibial Nerve Stimulation (PTNS) Therapy for Female Patients Suffering From Multiple Sclerosis
Brief Title: PTNS for Female Patients Suffering From Multiple Sclerosis
Acronym: PTNS-MS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Priya Padmanabhan, Fellowship Director, Female Pelvic Medicine and Reconstructive Surgery, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-168
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis; Overactive Bladder
Keywords: Multiple Sclerosis; MS; Overactive bladder; OAB
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, sham controlled.
Who Masked: Participant
Masking Description: Participant will be blinded to treatment group. Only the clinician providing the treatment will be aware of the treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active PTNS (Active Comparator): Once a week induction consisting of active PTNS treatments for 30 minutes for 12 consecutive weeks.
  Interventions: Device: PTNS Treatment
- Sham PTNS (Placebo Comparator): Once a week induction consisting of Sham PTNS treatments for 30 minutes for 12 consecutive weeks.
  Interventions: Device: Sham PTNS Treatment

INTERVENTIONS:
Device: PTNS Treatment — Patients will be placed in a comfortable position, sitting or supine. The treatment leg will be propped up comfortably on a footrest but draped and out of view from the patient. A 34-gauge needle electrode will be inserted at a 60-degree angle 5 cm cephalad to the medial malleolus and slightly posterior to the tibia. A PTNS surface electrode will be placed on the ipsilateral calcaneus as well as 2 inactive sham surface electrodes, 1 under the little toe and 1 on the top of the foot. When the PTNS lead set is connected to the Urgent PC stimulator, a current level of 0.5 to 9 mA at 20 Hz is selected based on each patient's foot and plantar motor and sensory responses. Treatment lasts 30 minutes and given once weekly for 12 consecutive weeks.
  Other Names: Urgent PC Neuromodulation System
  Arms: Active PTNS
Device: Sham PTNS Treatment — Patients will be positioned similarly as PTNS patients. A Streitberger needle will be used at the tibial nerve insertion site as described above to simulate needle placement. Three electrodes will be placed on the patient's foot, two active TENS electrodes and one inactive TENS electrode. The TENS "grounding pad" will be a gel electrode pad from a TENS unit device that is placed on the bottom of the foot just below the smallest toe. Another gel electrode will be placed on the top of the foot just above the small toe for conduction. These two electrodes will be connected to the TENS unit lead wires for sham stimulation. A third, inactive, gel electrode, will be placed near the medial aspect of the calcaneus to mimic the PTNS treatment. The TENS electrode will be connected by lead wires to the TENS unit set at 20 HZ. The TENS unit will be turned on and stimulation slowly increased to the patient's first sensory level and then turned off.
  Other Names: Biostim Transcutaneous electrical nerve stimulation (TENS) Unit
  Arms: Sham PTNS

SUMMARY:
This is a pilot, single blind, randomized, sham-controlled trial to assess the benefit of Percutaneous Tibial Nerve Stimulation (PTNS) in treating bladder overactivity (OAB) symptoms in multiple sclerosis (MS) patients. The data generated by this study would provide support for a future multi-institutional, randomized prospective trial.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, progressive inflammatory disorder of the central nervous system. It is caused by loss of myelin, the outer protective layer of the neuron, resulting in a disruption of the signal potentials that flow through the neurons. This can lead to a variety of sensory, visual, and motor disturbances. MS affects almost 1 million people in the United States with the prevalence being two to three times higher in women than in men. Over 80% of MS patients suffer from lower urinary tract symptoms, with OAB and urinary incontinence (UI) being the predominant bladder dysfunctions. OAB is characterized by sudden feeling of urgency, frequent urination, and urge incontinence. PTNS is an FDA approved treatment for OAB and is recommended as third line treatment for OAB by the American Urological Association (AUA) and Society of Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction (SUFU). However, it is not approved for MS and as such these treatments are not covered by insurance.

Here the investigators propose a pilot, double blind, randomized, sham-controlled trial to assess the benefit of PTNS in treating OAB symptoms in MS patients. The data generated by this study would provide support for a future multi-institutional, randomized prospective trial.

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis for Multiple Sclerosis (Clinically isolated syndrome (CIS), relapsing remitting (RRMS), secondary progressive (SPMS), and/or primary progressive (PPMS)), 18 years of age or older
* Self-reported bladder symptoms > 3 months
* Discontinued antimuscarinics/beta-3 agonists for > 2 weeks, and remain off for the duration of the study
* Capable of giving informed consent
* Ambulatory and able to use toilet independently without difficulty
* Capable and willing to follow all study-related procedures
* If of childbearing age, agree to practice approved birth-control methods (oral contraceptives, condom barrier, injection, diaphragm or cervical cap, vaginal contraceptive ring, intrauterine device (IUD), implantable contraceptive, surgical sterilization (bilateral tubal ligation), vasectomized partner(s))
* Subject agrees not to start any new treatments for urinary symptoms (medication or otherwise) during the treatment and follow-up periods.
* Subject agrees to maintain a stable dose on all current medications throughout the treatment and follow-up period.

Exclusion Criteria:

* Pregnant or planning to become pregnant during study duration
* Botox (BTX) use in bladder or pelvic floor muscles within past 6 months
* Pacemakers or implantable defibrillators
* Current urinary tract infection
* Active use of neuromodulation in any other form. If patient has InterStim, must be turned off for 2 weeks for a washout period and remain off during the entirety of the study.
* Current use of Transcutaneous Electrical Nerve Stimulation (TENS) in pelvic region, back or legs
* Previous PTNS treatment
* Participation in any clinical investigation involving or impacting gynecologic, urinary, or renal function within past 4 weeks

Note: For the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women assigned female at birth
Enrollment: 2 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Padmanabhan, MD, Principal Investigator — Beaumont Hospital, Royal Oak
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from December 2022 through December 2023.
Groups:
- Sham PTNS: Once a week induction consisting of Sham PTNS treatments for 30 minutes for 12 consecutive weeks.
  Sham PTNS Treatment: Patients will be positioned similarly as PTNS patients. A Streitberger needle will be used at the tibial nerve insertion site as described above to simulate needle placement. Three electrodes will be placed on the patient's foot, two active Urgent PC transcutaneous electrical nerve stimulation (TENS) electrodes and one inactive TENS electrode. The TENS "grounding pad" will be a gel electrode pad from a TENS unit device that is placed on the bottom of the foot just below the smallest toe. Another gel electrode will be placed on the top of the foot just above the small toe for conduction. These two electrodes will be connected to the TENS unit lead wires for sham stimulation. A third, inactive, gel electrode, will be placed near the medial aspect of the calcaneus to mimic the PTNS treatment. The TENS electrode will be connected by lead wires to the TENS unit set at 20 HZ. The TENS unit will be turned on and stimulation slowly increased to the patient's first sensory level and then turned off.
Period: Overall Study
Arm/Group | Active PTNS | Sham PTNS
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were zero patients randomized to the sham PTNS group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active PTNS | Sham PTNS | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) |  | 47 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: The Overall Patient Reported Change of Bladder Overactivity (OAB) Symptoms in MS Patients as Reported on the Patient Global Impression of Improvement (PGI-I) Questionnaire
Description: The PGI-I is a self-reported measure of symptom change after treatment completion. This is a validated 1-question tool. Subjects score their urinary condition now compared to how it was before starting treatment. The score ranges from 1-7. 1= very much better, 2 = much better, 3 = a little better, 4=no change, 5= a little worse, 6= much worse, 7 = very much worse. A higher score indicates a worse outcome. Only one participant completed the primary outcome, thus that subject score will be reported.
Time Frame: One week after completing all 12 treatments
Population: Of the 2 patients enrolled, only 1 patient completed the study and the primary outcome measure. The other subject withdrew prior to the primary outcome measure.
Measure: Number; unit: score
Arm/Group | Active PTNS | Sham PTNS
Number analyzed (Participants) | 1 | 0
score | 4 |

2. Secondary Outcome: Change in Urinary Voids in Response to the Treatment Using a 3-day Voiding Diary
Description: Study participants will complete a 3-day voiding diary to record number of voids. Investigators will analyze the change in urinary voids from before to after treatment. A positive number indicates more voids, and a negative number indicates fewer voids.
Time Frame: At baseline and one week after completing all 12 treatments, Visit 13
Population: Of the 2 patients enrolled, only 1 patient completed the study and the secondary outcome measure. The other subject withdrew prior to the secondary outcome measure.
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Active PTNS | Sham PTNS
Number analyzed (Participants) | 1 | 0
number of voids | 1 (0) |

3. Secondary Outcome: Change in Urinary Incontinence Episodes in Response to the Treatment Using a 3-day Voiding Diary
Description: Study participants will complete a 3-day voiding diary to record number of urinary incontinence episodes over a 3-day period. Investigators will analyze the change in urinary incontinence episodes from before to after treatment. A positive number indicates more episodes, and a negative number indicates fewer episodes.
Time Frame: At baseline and one week after completing all 12 treatments, Visit 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of urgency incontinence episodes
Arm/Group | Active PTNS | Sham PTNS
Number analyzed (Participants) | 1 | 0
number of urgency incontinence episodes | -3 (0) |

4. Secondary Outcome: Change in Urinary Urgency Episodes in Response to the Treatment Using a 3-day Voiding Diary
Description: Study participants will complete a 3-day voiding diary to record the number of urgency episodes over a 3-day period. Investigators will analyze the change in urinary urgency episodes from before to after treatment. A positive number indicates more episodes, and a negative number indicates fewer episodes.
Time Frame: At baseline and one week after completing all 12 treatments, Visit 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of urgency episodes
Arm/Group | Active PTNS | Sham PTNS
Number analyzed (Participants) | 1 | 0
number of urgency episodes | 1 (0) |

5. Secondary Outcome: Change in Overactive Bladder Symptoms in Response to the Treatment Using the Overactive Bladder Quality of Life Short Form Questionnaire.
Description: The Overactive Bladder quality of life questionnaire measures the impact of PTNS treatment on patient quality of life. Patients score symptom severity and impact on quality of life on a scale 1-6, with 1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit, 5=a great deal, and 6=a very great deal. Symptom severity raw score is calculated from questions 1-6; the lowest possible raw score is 6, the highest score is 36. The health-related quality of life (HRQL) raw score is calculated similarly from questions 1-13; the lowest possible score is 13 and highest score is 78. The formula (actual raw score - lowest possible raw score)/highest possible raw score times 100 is applied to each raw score, which are added to give a final score in the range 0 to 166.6, with low scores indicating fewer symptoms and impact, and high scores indicating more symptoms and impact. Change from baseline is reported, with a positive number indicating worsening and a negative number indicating improvement.
Time Frame: At baseline and one week after completing all 12 treatments, Visit 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PTNS | Sham PTNS
Number analyzed (Participants) | 1 | 0
score on a scale | -47.69 (0) |

ADVERSE EVENTS:
Time Frame: Approximately 14 weeks
Description: Adverse event monitoring occurred between start of treatment to the end of study participation, approximately 14 weeks including the last follow-up visit.
Arm/Group | Active PTNS | Sham PTNS
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Recruiting challenges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT05422625/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05422625/ICF_001.pdf